CLINICAL TRIAL: NCT01646736
Title: Evaluation of Efficacy and Safety of Glucocorticosteroid Combined With Oral T2 (Chloroform/Methanol Extract of Tripterygium Wilfordii Hook F) in the Treatment of Patients With Lupus Nephritis.
Brief Title: Efficacy and Safety of Tripterygium Wilfordii in Patients With Lupus Nephritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Fengchun Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T2WILN
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Nephritis, Lupus
Keywords: Lupus Nephritis; Cyclophosphamide; Tripterygium
MeSH Terms: conditions — Lupus Nephritis | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GC+CYC (Placebo Comparator): Patients were treated with Glucocorticosteroid and Cyclophosphamide.
  Interventions: Drug: Cyclophosphamide; Drug: GC
- GC+T2 (Experimental): Patients were treated with Glucocorticosteroid and oral T2 (chloroform/methanol extract of Tripterygium wilfordii Hook F).
  Interventions: Drug: Tripterygium wilfordii Hook F; Drug: GC

INTERVENTIONS:
Drug: Tripterygium wilfordii Hook F — Oral T2(Tripterygium wilfordii Hook F) 20mg thrice daily for 24 weeks.
  Arms: GC+T2
Drug: Cyclophosphamide — Cyclophosphamide 1.0 intravenous every month.
  Arms: GC+CYC
Drug: GC — Prednisone or equivalent 1 mg/kg/d(up to 60 mg), gradually tapering to 7.5mg/d in 24 weeks.

SUMMARY:
Evaluation the clinical efficacy and safety profile of glucocorticosteroid combined with oral T2 (chloroform/methanol extract of Tripterygium wilfordii Hook F) in the treatment of patients with lupus nephritis. Open-labeled, randomized, prospective multi-center clinical trial. Observation period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years with informed consent
* SLE defined by meeting 4 or more ACR classification criteria
* Biopsy-proven active proliferative lupus glomerulonephritis ISN classification Class III or IV
* Active renal disease

Exclusion Criteria:

* Pregnant, lactating or further fertility requirements
* Serum creatinine > 3 mg/dL
* Serum ALT or AST > 3 times upper limit of normal
* Severe, progressive renal, hepatic, hematological, gastrointestinal, pulmonary, cardiovascular, neurological, endocrine or cerebral disease
* Previous treated with cyclophosphamide or T2.
* Not discontinuing MMF, azathioprine, leflunomide, methotrexate, calcineurin inhibitor before 1 month of randomization.
* Active or chronic infection, including HIV, HCV, HBV, tuberculosis
* Patient with malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Renal Response | 24 weeks.
  The proportion of patients achieving Complete Response (CR) and Partial Response(PR).

SECONDARY OUTCOMES:
Renal Function | 24 weeks
  The change in glomerular filtration rate(GFR) from baseline to week 24.
Serum Albumin Level | 24 weeks
  The change in serum albumin level from baseline to week 24.
Complement | 24 weeks
  The change in complement components from baseline to week 24, including: CH50(total complement activity), C3 and C4 level measured by nephelometry.
Anti-dsDNA | 24 weeks
  The change in anti-dsDNA antibody titers from baseline to week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Fengchun Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Deptment of Rheumatology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China